CLINICAL TRIAL: NCT05653778
Title: Scrambler Therapy for Corticobasal Syndrome-Associated Pain
Acronym: ST-CBS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00343996
Record Dates: First submitted 2022-11-29; First posted 2022-12-16 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Corticobasal Degeneration; Corticobasal Syndrome; Pain, Neuropathic
Keywords: Corticobasal Degeneration; scrambler therapy; Corticobasal syndrome; neuropathic pain; neuropathy
MeSH Terms: conditions — Corticobasal Degeneration; Neuralgia

STUDY DESIGN:
Intervention Model Description: Randomly assigned scrambler therapy or TENS treatment to patients.
Who Masked: Participant
Masking Description: Patients will be masked on whether they will receive scrambler therapy or TENS treatment for neuropathic pain.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Scrambler therapy (Experimental): Scrambler Therapy is a non-invasive neuromodulation approach using superficial electrocardiogram (ECG) electrodes in paired channels on the involved dermatomes to send "non-pain" information along the existing nerve pathways, which can modify peripheral and central sensitization.
  Interventions: Device: Scrambler therapy
- TENS treatment (Active Comparator): Transcutaneous electrical nerve stimulation (TENS) is a battery-powered device which delivers low-voltage electrical current through superficial electrocardiogram (ECG) electrodes placed on the surface of the skin to provide pain relief.
  Interventions: Device: TENS treatment

INTERVENTIONS:
Device: Scrambler therapy — Superficial electrocardiogram (ECG) electrodes are placed on the dermatomes involved with pain, above the area of pain itself. Each treatment lasts 30-40 minutes or until pain relief is obtained.
  Arms: Scrambler therapy
Device: TENS treatment — Superficial electrocardiogram (ECG) electrodes are placed on the dermatomes involved with pain, above the area of pain itself. Each treatment lasts 30-40 minutes or until pain relief is obtained.
  Arms: TENS treatment

SUMMARY:
The goal of this pilot trial is to test whether scrambler therapy (ST) is an effective treatment for neuropathic pain in patients with corticobasal syndrome (CBS).

The main question it aims to answer is:

Will ST reduce pain scores by at least 33% at one month in this pilot trial, justifying further multi-center trials?

Participants will:

* be randomly assigned treatment from either transcutaneous electrical nerve stimulation (TENS) or ST for pain initially (eventually all patients will receive ST).
* have superficial electrocardiogram (ECG) electrodes placed on the dermatomes involved with pain
* obtain treatment lasting 30-40 minutes or until pain relief is obtained

Researchers will compare patient's response to pain relief with TENS and ST to determine if ST is an effective treatment for central neuropathic pain.

DETAILED DESCRIPTION:
Pain can be a common non-motor complication of corticobasal syndrome (CBS), which is a rare debilitating parkinsonian disorder that lacks disease-modifying therapies. Pain in CBS typically increases in severity as the disease progresses and adversely impacts quality of life (including sleep and daily function). Scrambler therapy is a non-invasive electrical approach to neuromodulation that sends "nonpain" information along the existing nerve pathways to modify peripheral and central sensitization with success in randomized controlled trials treating such difficult neuropathies as spinal cord stenosis, post-herpetic neuropathy and failed back syndrome; chemotherapy induced neuropathy; and neuromyelitis optica spectrum disorder (NMOSD). To date, four patients with CBS treated empirically with ST have experienced long lasting pain relief with treatment, suggesting a novel approach to a vexing symptom.

An estimated 35-80% of patients with Parkinson disease experience pain and it is highly likely that pain is more frequent in CBS, though estimates are lacking because CBS is a rare syndrome. This pain can be related to dystonia, musculoskeletal, radicular-peripheral neuropathic, and central neuropathic pain syndromes. Similar symptoms are found in patients with CBS. Currently, there are no FDA approved disease-modifying treatments. Although treatments for pain have been helpful, ultimately adjunct therapies are needed as the disease progresses. A simple, low-cost, non-invasive available treatment to reduce the pain of CBS is sorely needed. This pilot trial will provide data on which to design a larger randomized controlled trial.

Research Hypothesis: Scrambler Therapy (ST) will reduce pain scores by at least 33% at one month in this pilot trial, justifying further multi-center trials.

ELIGIBILITY:
Inclusion Criteria:

* men and women, ≥50 years of age or older with CBS with an average daily pain rating of > 4 out of 10, using the following question from the Brief Pain Inventory: "Please rate your pain by circling the one number that best describes your (abdominal) pain/discomfort on average over the past week. (Scale 0-10; 0= No pain, 10= Pain as bad as you can imagine)
* English speakers or English proficiency
* They must have a life expectancy > 90 days per their treating neurologist.
* The patient must be able to understand the study regimen, its requirements, risks, and discomforts, and is able and willing to sign an informed consent form.

Exclusion Criteria:

* Pregnant women, nursing women, women of childbearing potential or their sexual partners who are unwilling to employ adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device, surgical sterilization, subcutaneous implants, abstinence, etc.). Other exclusions include the following:
* Use of an investigational agent for pain control concurrently or within the past 30 days,
* History of an allergic reaction or previous intolerance to transcutaneous electronic nerve stimulation;
* Patients with implantable drug delivery systems, e.g. Medtronic Synchromed, baclofen pumps.
* Patients with heart stents or metal implants such as pacemakers, automatic defibrillators, cochlear implants, aneurysm clips, vena cava clips and skull plates. (Metal implants for orthopedic repair, e.g. pins, clips, plates, cages, joint replacements are allowed).
* Medical exclusions include: patients with a history of myocardial infarction or ischemic heart disease within the past six months; patients with history of epilepsy, brain damage, or symptomatic brain metastases; skin conditions such as open sores that would prevent proper application of the electrodes; or other medical or other condition(s) that in the opinion of the investigators might compromise the objectives of the study.

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Change in patient-reported average daily pain using the Modified Brief Pain Index | Day 0 to Day 30 and 90
  The primary objective is to determine the change in patient-reported average daily pain from Day 0 to Day 30 and 90 as measured on a numerical scale of 0-10 (0=no pain; 10=worst pain in life) using the Modified Brief Pain Index.

SECONDARY OUTCOMES:
Change in patient-reported Global Impression of Change (PGIC) | Day 0, Day 30 and Day 90
  Changes in the Patient Global Impression of Change score 1 to 7 with 1 representing no change and 7 representing "a great deal better"

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Pantelyat, MD, Principal Investigator — Department of Neurology, Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No